CLINICAL TRIAL: NCT06883162
Title: Randomized Controlled Trial of Varenicline to Treat Tobacco and Cannabis Co-Use (RECLAIM)
Brief Title: Cannabis-Tobacco Co-Use Treatment Study
Acronym: RECLAIM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erin McClure, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00136115; R01CA290842 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use Disorder; Tobacco Use Cessation; Cannabis Use; Cannabis Use Disorder; Marijuana Use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Marijuana Use | interventions — Varenicline; Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline (Experimental): Participants will be randomized 1:1 to varenicline or matched placebo. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1 mg b.i.d. starting on Day 8. Dosing of 2 mg per day will be maintained for the next 11 weeks.
  Interventions: Drug: Varenicline; Behavioral: Counseling; Behavioral: Psychosocial modules
- Placebo (Placebo Comparator): Participants will be randomized 1:1 to varenicline or matched placebo.
  Interventions: Behavioral: Counseling; Behavioral: Psychosocial modules

INTERVENTIONS:
Drug: Varenicline — Participants will be randomized 1:1 to varenicline or matched placebo. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1 mg b.i.d. starting on Day 8. Dosing of 2 mg per day will be maintained for the next 11 weeks.
  Arms: Varenicline
Behavioral: Counseling — Research staff will provide skills-based counseling at weekly visits. Weekly counseling sessions will include discussion of online intervention modules, while providing skills-based strategies focused on enlisting social support, recognizing triggers, managing craving/withdrawal/stress, etc. Staff will use motivational enhancement techniques to address tobacco cessation, cannabis reduction or abstinence, and medication adherence.
Behavioral: Psychosocial modules — Participants will have access to online modules addressing tobacco and cannabis co-use to support cessation and/or reduction. Content includes 12 virtual modules combining cognitive behavioral therapy (CBT) and motivational enhancement (MET) to address tobacco, cannabis, and their co-use.

SUMMARY:
The purpose of the RECLAIM study is to evaluate the effectiveness of varenicline (sometimes known as Chantix) compared to placebo (an inactive substance) for the treatment of cigarettes and cannabis (marijuana). Varenicline is not FDA approved for the combination treatment of cigarette abstinence and cannabis reduction or abstinence. All participants will also receive counseling and access to online treatment modules during a quit attempt for cigarettes and a reduction attempt for cannabis. This study is being conducted by the Medical University of South Carolina. All procedures are conducted remotely and there is no in-person visits are needed.

To qualify, participants must be 18 or older, live in South Carolina, use cigarettes and cannabis, and are interested in quitting cigarettes and reducing cannabis.

DETAILED DESCRIPTION:
Tobacco-cannabis co-use results in established harms, yet there are currently no recommended treatment strategies for co-use. The scientific premise of this proposal is based on work conducted by our group demonstrating that: 1) cannabis co-use adversely impacts cigarette abstinence and those co-using cannabis have nearly double the odds of tobacco treatment failure, 2) varenicline may be efficacious in treating CUD, and 3) cannabis reduction (vs. abstinence) may be a potentially more appealing treatment goal. Therefore, this project proposes to evaluate varenicline versus placebo on cigarette abstinence and cannabis use reduction or abstinence among adults who co-use. To bolster outcomes, both groups will receive an evidence-based psychosocial intervention that includes real-time and asynchronously delivered content (all delivered virtually), that leverages the co-use intervention used by Budney (Consultant) as well brief weekly counseling and check-in sessions that we have used in previous and ongoing studies. Asynchronous content (web-based modules) is standardized and through a tailored approach to counseling, the intervention will allow for participant preference for cannabis reduction or abstinence. The selection of this combination treatment for tobacco-cannabis co-use is based on rigorous prior research demonstrating: 1) efficacy of varenicline for tobacco cessation, 2) preliminary efficacy of varenicline for cannabis use, and 3) acceptable, psychosocial co-use treatment modules that have the potential to augment a robust pharmacotherapy to improve outcomes.

Investigators propose a completely remote 12-week treatment trial among adults in South Carolina (ages 18+; N=200) who co-use cigarettes and cannabis regularly. Participants will be included who smoke cigarettes daily or near daily (20+ days in the past 30) and have used cannabis at least 3 times per week in the past month. Participants will be randomized 1:1 to varenicline or placebo and all participants will receive the platform psychosocial intervention. The aims of the study are to: 1) evaluate rates of 7-day biochemically confirmed point prevalence abstinence (PPA) from cigarettes at the 12-week EOT visit comparing varenicline + psychosocial intervention to the placebo + psychosocial intervention participants (Aim 1), 2) compare cannabis use frequency and amount between varenicline and placebo groups during treatment (Weeks 1-12; Aim 2), and 3) explore differential treatment outcomes among male vs. female participants (Exploratory Aim).

ELIGIBILITY:
Inclusion criteria:

1. Ages 18 and over (no upper age limit)
2. Must smoke at least 5 tobacco cigarettes per day on at least 20 out of the past 30 days for the past 3 months
3. Must express interest in quitting tobacco
4. Must express interest in cannabis reduction and/or cessation
5. Must submit a positive instant-read test for cotinine and cannabis prior to enrollment
6. Must self-report cannabis use (THC-dominant products) on at 3 days per week out of the past 30 days
7. Must be willing to take varenicline or placebo for 12 weeks
8. Must reside in South Carolina

Exclusion criteria:

1. Any significant or acutely unstable medical, psychiatric, or substance use problem (including clinically significant disorders) that would contraindicate research, interfere with safety, compromise data integrity, or preclude consistent study participation
2. Pregnant or trying to become pregnant
3. Use of medications with smoking cessation efficacy
4. Regular use of e-cigarettes or other tobacco products (<10 days in the past month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Cigarette abstinence | Final 7 days of treatment (Week 11 through Week 12)
  Biochemically-confirmed 7-day point prevalence abstinence from tobacco

SECONDARY OUTCOMES:
Changes in cannabis use frequency | Weeks 1 through 12 of treatment
  Assess changes in cannabis using days (frequency) during treatment
Changes in cannabis use amount | Weeks 1 through 12 of treatment
  Assess changes in sessions (episodes) of cannabis use per day (amount) during treatment

OTHER OUTCOMES:
Sex differences in tobacco and cannabis outcomes | Weeks 1 through 12 of treatment
  Biochemically-confirmed 7-day point prevalence abstinence from tobacco, cannabis use days and sessions of cannabis use per day

CONTACTS AND LOCATIONS:
Overall Officials: Erin Mcclure, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina - Charleston, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A final de-identified data set will be made available for retrieval and analysis of secondary outcomes, upon request to the Principal Investigator.